CLINICAL TRIAL: NCT01260597
Title: Re-engagement in Evidence-based Quit Line Treatment for Low Income Smokers
Brief Title: Tobacco Quit Line Re-enrollments for the Underserved
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consumer Wellness Solutions (Industry)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0002; 1R21CA14156801 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Smoking
Keywords: smoking; quit line re-enrollment and IVR systems
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Life Style Counseling (Experimental): For individuals who report being quit, a brief congratulatory message will be delivered, independent of each arm of the study they were randomized to. For individuals who report not being quit and are randomized to the intervention condition, tailored messages are delivered via the IVR system. The automated calls would include an assessment of the individual's interest in another quit attempt and deliver brief, tailored messages to perceived barriers for re-engaging into treatment. The system is programmed to transfer the caller to a live quit line counselor if the individual is willing to re-engage in cessation treatment.
  Interventions: Behavioral: IVR intervention
- Life Counseling (Active Comparator): For individuals who report being quit, a brief congratulatory message will be delivered, independent of each arm of the study they were randomized to. For individuals who report still smoking the IVR will thank them for their time and the call will end.
  Interventions: Behavioral: IVR control

INTERVENTIONS:
Behavioral: IVR intervention — If individuals report having any smoking in the previous 30 days, the IVR will deliver questions to identify barriers to quit line re-enrollment and motivational messages to promote the re-enrollment
  Arms: Life Style Counseling
Behavioral: IVR control — If individuals report any smoking in the last 30 days the IVR will thank them for their time and the call will end
  Arms: Life Counseling

SUMMARY:
The purpose of this proposed study is to develop, refine and test the use of Interactive Voice Response (IVR) technology as a means of increasing re-engagement of low income smokers in telephone support for tobacco cessation (quit lines). If this strategy proves to be acceptable and feasible, it may offer a technological solution to increase access to and utilization of a widely available evidence-based form of behavioral treatment for low income smokers.

The primary aims of this research are to:

1. Develop an IVR system that delivers tailored audio messages to increase low income smokers' re-engagement in treatment offered by two state quit lines (Washington and Indiana). The investigators will develop: a) a menu of audio messages that can be delivered by an IVR system; b) an IVR algorithm (i.e., a set of decision rules) to make proactive automated calls to deliver brief, tailored messages for re-engaging low income smokers who previously used the quit line.
2. Evaluate the feasibility and efficacy of an IVR system as a tool to re-engage low income smokers into quit line treatment measured by number of IVR calls answered, number of smokers who re-engage in treatment and satisfaction with IVR calls. Hypothesis 2.1 - It is hypothesized that the rates of re-engagement into treatment among those receiving the IVR intervention will be higher than smokers not proactively invited to re-engage in quit line services.

DETAILED DESCRIPTION:
We propose a randomized controlled trial to compare re-engagement into quit line treatment between low income smokers receiving IVR intervention to re-engage into treatment through quit line services and those receiving usual care (no intervention to re-engage). Subjects will be recruited from two state quit lines (Washington (WA) and Indiana (IN)). WA and IN were selected because they both contract with Free & Clear for quit line services and have supported research collaborations in the past. Both states have agreed to participate in this study. Three thousand subjects will be randomized to the intervention or usual care prior to entry into the IVR calling database. This sampling frame was defined based in our past research experience in using similar method to re-engage low income smokers from ethnic populations and assumed a high proportion of invalid phone numbers and difficulties on successfully reaching individuals even after several call attempts. In our previous re-engagement study, 29% of the phone numbers provided by quit line users were invalid 12 months later and 38% of the subjects were never reached after five attempted calls. Therefore, in this study we are anticipating successfully reaching 30% of the sample.

This is a feasibility study and the main outcome is re-engagement into treatment, measured by re-enrollment into quit line support after receiving the IVR intervention. Process measures are IVR calls answered and satisfaction with IVR calls. Thirty-day point prevalence abstinence at 6 months after intervention will be also measured, as a way to preliminarily evaluate the efficacy of this intervention.

The target population of this study is low income smokers, defined as being a Medicaid recipient or uninsured by the time of their first enrollment into quit line treatment. This working definition for eligibility criterion was chosen because health insurance status is routinely assessed in the provision of quit line services and it is a good proxy indicator of income.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Medicaid or uninsured, 18 years or older, able to read and speak English, provided verbal consent to be contacted by quit line to follow-up, sought quit line services for being primarily a smoker

Exclusion Criteria:

* Primary use of other forms of tobacco such as smokeless tobacco, not understanding English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2985 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Quit line re-enrollment | At 6 months
  Evaluate the feasibility and efficacy of an IVR system as a tool to re-engage low income smokers into quit line treatment measured by number of IVR calls answered, number of smokers who re-engage in treatment and satisfaction with IVR calls.

SECONDARY OUTCOMES:
Tobacco Abstinence | At 6 months
  Thirty-day point prevalence abstinence at 6 months after intervention will be also measured, as a way to preliminarily evaluate the efficacy of this intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Carlini, PhD, MPH, Principal Investigator — Free & Clear, Inc.
Locations (1):
- Free & Clear, Inc, Seattle, Washington, United States

REFERENCES:
- [Derived] Carlini BH, McDaniel AM, Weaver MT, Kauffman RM, Cerutti B, Stratton RM, Zbikowski SM. Reaching out, inviting back: using Interactive voice response (IVR) technology to recycle relapsed smokers back to Quitline treatment--a randomized controlled trial. BMC Public Health. 2012 Jul 6;12:507. doi: 10.1186/1471-2458-12-507. PMID 22768793